CLINICAL TRIAL: NCT02679300
Title: The Influence of a Virtual Reality Environment on Pain Perception During Exercises for Patients With Chronic Non-specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Virtual Reality and Pain Perception During Exercises for Patients With Chronic Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Thomas Matheve, PT, MSc, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TMatheveVR&Pain
Record Dates: First submitted 2016-02-04; First posted 2016-02-10 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Virtual Reality; Serious Gaming; Exercise Therapy; Distraction
MeSH Terms: interventions — Control Groups

ARMS (2):
- Virtual reality group (Experimental): During a single intervention session, participants will perform 2 sets of 2 minutes of pelvic tilt exercises using serious games. These serious games have to be controlled by pelvic tilts. Patients will perform the exercises in a standing position in front a TV-screen, on which the games will be displayed. Wireless motion sensors will be mounted to the patient's spine and pelvis to track the movements of the pelvis.
  Interventions: Other: Virtual reality exercise group
- Control group (Active Comparator): During a single session intervention, participants will perform 2 sets of 2 minutes of pelvic tilt exercises without a serious game. Patients will perform the exercises in a standing position. The number of repetitions and the tempo of the pelvic tilts will be indicated using a metronome.
  Interventions: Other: Conventional exercise group (control group)

INTERVENTIONS:
Other: Virtual reality exercise group
  Arms: Virtual reality group
Other: Conventional exercise group (control group)
  Arms: Control group

SUMMARY:
Immersion in a virtual reality environment has been shown to reduce pain during a variety of painful medical procedures, such as wound care for burn patients and dental care. Often, serious games are used to distract patients from this painful procedures. Recently, serious games have also been developed for patients with low back pain. Because patients with low back pain frequently experience pain during exercises, the investigators hypothesize that exercising with serious games can reduce the pain intensity and the time spent thinking of pain during exercises. To test this hypothesis, the investigators will conduct a randomized controlled trial where two groups will be compared: the experimental group will perform one session of exercises with serious games, while the control group will perform one session of the same exercises without the serious games.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific low back pain, with or without referred pain to the legs
* Age 18-65
* Able to understand Dutch
* A minimum pain intensity of 3/10 on the numeric pain rating scale at the time of the test
* Being familiar with pelvic tilt exercises

Exclusion Criteria:

* Spinal surgery in the past
* Pregnancy
* Serious underlying pathologies (e.g. multiple sclerosis, tumors,…)
* Signs or symptoms of nerve root involvement
* Known skin-allergy for tape

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Average pain intensity during exercises using the numeric pain rating scale | Day 1
  Immediately after the intervention, patients will be asked to indicate the average pain they experienced during the exercises using the numeric pain rating scale (0-10)
Time spent thinking of the pain using a numeric rating scale | Day 1
  Immediately after the intervention, patients will be asked to indicate the average time they spent thinking of their pain during the exercises using a numeric rating scale ranging from 0 ("not at all") to 10 ("all the time")

SECONDARY OUTCOMES:
Pain intensity after the exercises using a numeric rating scale | Day 1
  Patients will be asked to indicate their pain immediately after the exercises using the numeric pain rating scale (0-10)
Harmfulness of the exercises using a numeric rating scale | Day 1
  Immediately after the intervention, patients will be asked to indicate how harmful they thought the exercises were for their lumbar spine on a numeric rating scale ranging from 0 ("not harmful at all") to 10 ("extremely harmful").

OTHER OUTCOMES:
Number of pelvic tilts | Day 1
  During the exercises the pelvis and lumbar spine of the participants will be recorded with a digital videocamera to capture the number of pelvic tilts during the exercises. This outcome measure will primarily be used as possible covariate
Immersion (questionnaire will be used to measure the level of immersion) | Day 1
  Immediately after the intervention, the immersive experience questionnaire will be used to measure the level of immersion

CONTACTS AND LOCATIONS:
Locations (1):
- Hasselt University, Hasselt, Belgium

REFERENCES:
- [Derived] Matheve T, Bogaerts K, Timmermans A. Virtual reality distraction induces hypoalgesia in patients with chronic low back pain: a randomized controlled trial. J Neuroeng Rehabil. 2020 Apr 22;17(1):55. doi: 10.1186/s12984-020-00688-0. PMID 32321516